CLINICAL TRIAL: NCT01696240
Title: Udenafil Therapy to Improve Symptomatology, Exercise Tolerance and Hemodynamics in Patients With Mild Pulmonary Hypertension [ULTIMATE-Mild PHT]
Brief Title: A Randomized Trial of Udenafil Therapy in Patients With Mild Pulmonary Hypertension [ULTIMATE-Mild PHT]
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yong-Jin Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1202-005-396
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Mild Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Exercise Capacity; Cardiopulmonary Exercise Test; Udenafil (Zydena); Phosphodiesterase Type 5 Inhibitors
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Capsule that is identically appearing with udenafil will be administered to patients in placebo group. For the first 4 weeks, patients will receive 50 mg of placebo drug two times a day, and then the dosage will be doubled to 100 mg two times a day for next 8 weeks.
  Interventions: Drug: Placebo
- Udenafil (Active Comparator): Patients will receive 50 mg of udenafil two times a day, and then the dosage will be doubled to 100 mg two times a day for next 8 weeks.
  Interventions: Drug: Udenafil (Zydena)

INTERVENTIONS:
Drug: Placebo — Capsule, appears identical with udenafil, will be provided by Dong-A pharmaceutical company. Patients will receive 50 mg of placebo drug two times a day for 4 weeks, and then the dosage will be escalated to 100 mg two times a day for next 8 weeks.
  Other Names: The same placebo drug of NCT01553721.
  Arms: Placebo
Drug: Udenafil (Zydena) — Udenafil (Zydena), a newly developed PDE-5 inhibitor by Dong-A pharmaceutical company, will be administered to patients in this group, 50 mg two times a day for 4 weeks, and then the dosage will be escalated to 100 mg two times a day for next 8 weeks.
  Other Names: DA-8159 (CAS No 268203-93-6)
  Arms: Udenafil

SUMMARY:
The investigators hypothesized that udenafil, a newly developed phosphodiesterase type 5 inhibitor, would improve symptom, exercise capacity and hemodynamic status in patients with mild pulmonary hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is a devastating progressive disease increasingly debilitating symptoms. In the past few years, treatment of pulmonary hypertension has undergone an extraordinary evolution. A selective PDE-5 inhibitor, Sildenafil, has been shown to be as an effective pulmonary vasodilator as inhaled NO in patients with primary pulmonary hypertension and has recently been shown to improve exercise capacity, resting hemodynamics, and WHO functional class in patients with pulmonary hypertension. However, to date, the effect of Sildenafil have been mainly studied in patients with advanced disease.

Udenafil (Zydena), a newly developed PDE-5 inhibitor, has been proved to have similar efficacy and safety profile, compared with other PDE-5 inhibitors. However, to date, the effect of Udenafil in mild pulmonary HT has never been evaluated. Therefore, we hypothesized that Udenafil, a newly developed phosphodiesterase type 5 inhibitor, would improve symptom, exercise capacity and hemodynamic status in patients with mild pulmonary hypertension.

In this 12-week, randomized, double-blind, placebo-controlled trial, patients with mild pulmonary hypertension will be enrolled according to the eligibility criteria. After randomization, study participants will be assigned to receive either 50mg of Udenafil or placebo two times a day for 4 weeks, and then the dosage will be doubled to 100mg two times a day for next 8 weeks. Participants will attend study visits at baseline and weeks 4 and 12. Physical examination, medical history review, blood sample collection and electrocardiogram will be conducted on each study visits. At baseline and week 12, participants will undergo cardiopulmonary exercise test and exercise echocardiography. At every study visits, researchers will collect health information.

ELIGIBILITY:
Inclusion Criteria:

- Mild pulmonary hypertension defined as estimated pulmonary arterial systolic pressure of 30-50 mmHg (TR jet velocity of 2.5-3.4 m/sec) with current New York Heart association (NYHA) class II-IV symptoms, left ventricular ejection fraction (LVEF) greater than or equal to 50% at the time of study entry

Exclusion Criteria:

* Hospitalization for decompensated heart failure or acute treatment with intravenous loop diuretics or hemofiltration in the 12 months before study entry
* E/E' ratio greater than or equal to 15 measured by echocardiography
* E/E' ratio greater than or equal to 8, and left atrial volume index (LAVI) greater than or equal to 40 ml/m2 measured by echocardiography
* E/E' ratio greater than or equal to 8 measured by echocardiography, and plasma BNP concentration greater or equal to 200 pg/ml
* Significant obstructive or restrictive lung disease
* Valve disease (greater than mild stenosis or regurgitation)
* Hypertrophic cardiomyopathy
* Infiltrative or inflammatory myocardial disease
* Pericardial disease
* Primary pulmonary arteriopathy
* Has neuromuscular, orthopedic, or other non-cardiac condition that prevents individual from exercise testing
* Has experienced myocardial infarction or unstable angina, or has undergone percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 60 days before study entry
* Non-cardiac illness with estimated life expectancy less than 1 year at the time of study entry, based on the judgment of the physician
* Current use of nitrate therapy
* Current use of other phosphodiesterase 5 inhibitors (ie. sildenafil, vardenafil, tadalafil) for treatment of impotence or pulmonary artery hypertension
* Current use of cytochrome P450 3A4 inhibitors (ie. ketoconazole, itraconazole, erythromycin, saquinavir, cimetidine, protease inhibitors for HIV)
* Severe hypotension (systolic blood pressure [SBP] less than 90mmHg or diastolic blood pressure [DBP] less than 50mmHg) or uncontrolled hypertension (SBP greater than 180mmHg or DBP greater than 100mmHg)
* Known severe renal dysfunction (estimated glomerular filtration rate [GFR] less than 30ml/min/1.73m2 by modified modification of diet in renal disease [MDRD] equation)
* Known severe liver disease (alanine transaminase [ALT] or aspartate aminotransferase [AST] level greater than three times the upper normal limit, alkaline phosphatase [ALP] or total bilirubin greater than two times the upper normal limit)
* History of leukemia, multiple myeloma or penile deformities that increase the risk for priapism (eg. Peyronie's disease)
* History of proliferative diabetic retinopathy, retinitis pigmentosa, nonischemic optic neuropathy, or unexplained visual disturbance
* Female patients currently pregnant or women of childbearing age who were not using contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change of maximal VO2 in cardiopulmonary exercise test | Baseline and 12th weeks
  Comparison between groups and within groups.

SECONDARY OUTCOMES:
Change of symptomatic status expressed as New York Heart Association (NYHA) functional class | Baseline, 4th week, and 12th week
  Comparison between groups and within groups.
Change of pulmonary artery systolic pressure (PASP) in echocardiography at rest and during exercise | Baseline and 12th week
  Comparison between groups and within groups.
Change of left ventricular systolic function expressed as ejection fraction (EF), fractional shortening (FS) in echocardiography | Baseline and 12th week
  Comparison between groups and within groups.
Change of ventilator efficiency (VE/VCO2 slope) in cardiopulmonary exercise test | Baseline and 12th week
  Comparison between groups and within groups.
Change of plasma concentration of BNP | Baseline, 4th week, and 12th week
  Comparison between groups and within groups.
All-cause death | 12th week
  The occurrence of all-cause mortality during 12 week follow-up
Cardiac death | 12th week
  The occurrence of cardiac death including sudden cardiac death during 12 week follow-up
Admission for heart failure | 12th week
  Admission due to congestive heart failure during 12 week follow-up
Composite clinical endpoints | 12th week
  Composite clinical endpoints during 12 week follow-up, are defined as follows:
  Composite of all-cause death and admission for heart failure Composite of cardiac death and admission for heart failure
Safety endpoint | 12th week
  Safety endpoint during 12 week follow-up, is defined as follows:
  Development of facial flushing, febrile sensation, eyeball pain, visual disturbance, headache, penile erection.
  Intolerance or development of other adverse drug reactions related with study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Jin Kim, MD, PhD, Study Chair — Seoul National University Hospital; Goo-Yeong Cho, MD, PhD, Principal Investigator — Seoul National University Hospital; Hyung-Kwan Kim, MD, PhD, Study Director — Seoul National University Hospital; Seung-Pyo Lee, MD, Study Director — Seoul National University Hospital; Yeonyee Yoon, MD, Study Director — Seoul National University Hospital; Kyung-Hee Kim, MD, Study Director — Seoul National University Hospital; In-Chang Hwang, MD, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] McLaughlin VV, Archer SL, Badesch DB, Barst RJ, Farber HW, Lindner JR, Mathier MA, McGoon MD, Park MH, Rosenson RS, Rubin LJ, Tapson VF, Varga J; American College of Cardiology Foundation Task Force on Expert Consensus Documents; American Heart Association; American College of Chest Physicians; American Thoracic Society, Inc; Pulmonary Hypertension Association. ACCF/AHA 2009 expert consensus document on pulmonary hypertension a report of the American College of Cardiology Foundation Task Force on Expert Consensus Documents and the American Heart Association developed in collaboration with the American College of Chest Physicians; American Thoracic Society, Inc.; and the Pulmonary Hypertension Association. J Am Coll Cardiol. 2009 Apr 28;53(17):1573-619. doi: 10.1016/j.jacc.2009.01.004. No abstract available. PMID 19389575
- [Background] National Pulmonary Hypertension Centres of the UK and Ireland. Consensus statement on the management of pulmonary hypertension in clinical practice in the UK and Ireland. Heart. 2008 Mar;94 Suppl 1:i1-41. doi: 10.1136/hrt.2007.132118. No abstract available. PMID 18276826
- [Background] Galie N, Hoeper MM, Humbert M, Torbicki A, Vachiery JL, Barbera JA, Beghetti M, Corris P, Gaine S, Gibbs JS, Gomez-Sanchez MA, Jondeau G, Klepetko W, Opitz C, Peacock A, Rubin L, Zellweger M, Simonneau G; ESC Committee for Practice Guidelines (CPG). Guidelines for the diagnosis and treatment of pulmonary hypertension: the Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS), endorsed by the International Society of Heart and Lung Transplantation (ISHLT). Eur Heart J. 2009 Oct;30(20):2493-537. doi: 10.1093/eurheartj/ehp297. Epub 2009 Aug 27. No abstract available. PMID 19713419
- [Background] Cheitlin MD, Hutter AM Jr, Brindis RG, Ganz P, Kaul S, Russell RO Jr, Zusman RM. Use of sildenafil (Viagra) in patients with cardiovascular disease. Technology and Practice Executive Committee. Circulation. 1999 Jan 5-12;99(1):168-77. doi: 10.1161/01.cir.99.1.168. No abstract available. PMID 9884398
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984
- [Background] Lewis GD, Shah R, Shahzad K, Camuso JM, Pappagianopoulos PP, Hung J, Tawakol A, Gerszten RE, Systrom DM, Bloch KD, Semigran MJ. Sildenafil improves exercise capacity and quality of life in patients with systolic heart failure and secondary pulmonary hypertension. Circulation. 2007 Oct 2;116(14):1555-62. doi: 10.1161/CIRCULATIONAHA.107.716373. Epub 2007 Sep 4. PMID 17785618
- [Background] Kim BH, Lim HS, Chung JY, Kim JR, Lim KS, Sohn DR, Cho JY, Yu KS, Shin SG, Paick JS, Jang IJ. Safety, tolerability and pharmacokinetics of udenafil, a novel PDE-5 inhibitor, in healthy young Korean subjects. Br J Clin Pharmacol. 2008 Jun;65(6):848-54. doi: 10.1111/j.1365-2125.2008.03107.x. Epub 2008 Mar 3. PMID 18318773
- [Background] Kang KK, Ahn GJ, Sohn YS, Ahn BO, Kim WB. DA-8159, a new PDE5 inhibitor, attenuates the development of compensatory right ventricular hypertrophy in a rat model of pulmonary hypertension. J Int Med Res. 2003 Nov-Dec;31(6):517-28. doi: 10.1177/147323000303100608. PMID 14708417